CLINICAL TRIAL: NCT01309334
Title: Pharmacoeconomic and Clinical Prospective Comparison of PET-scan and MRI in Patients With de Novo Multiple Myeloma Less Than 65 Years of Age Treated According to IFM/DFCI 2009 Clinical Trial.
Brief Title: Imaging Young Myeloma (IMAgerie JEune Myélome)
Acronym: IMAJEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STIC/10/03; 2010-A01382-37 (Other: Afssaps)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Myeloma
Keywords: MRI; PET-scan; multiple myeloma; prognosis; pharmacoeconomic analysis
MeSH Terms: conditions — Multiple Myeloma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PET scan — Performed at diagnosis, after 3 cycles of induction therapy, and at completion of therapy
Procedure: MRI — Performed at diagnosis, after 3 cycles of induction therapy, and at completion of therapy

SUMMARY:
Multicenter open-label prospective comparative study of PET-scan and MRI at the time of diagnosis, after 3 cycles of induction therapy (RVD) and at the completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic de novo multiple myeloma
* less than 65 years of age
* enrolled in the IFM/DFCI clinical trial

Exclusion Criteria:

* 66 years of age or more
* not eligible for high-dose therapy
* Cons-indications to MRI or PET-Scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least one lesion not detected on the MRI lesions | At diagnosis

SECONDARY OUTCOMES:
Negativity of the exam after 3 cycles of chemotherapy and just before the maintenance treatment | 3 months and 7 months
Number of lesions at diagnosis | Inclusion (diagnosis)
diffuse disease at diagnosis | Diagnosis time (inclusion)
Direct costs of PET and MRI at diagnosis, after the first cycles of chemotherapy and before the maintenance treatment | Inclusion, 3 months and 7 months

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital "CHU du Morvan", Brest
  - Hospital "Côte de Nacre", Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital "Hôpital Michallon", Grenoble
  - Le Mans Hospital, Le Mans
  - Lille University Hospital "Claude Huriez", Lille
  - Lyon University Hospital, Lyon
  - "Institut Paoli Calmettes", Marseille
  - Metz University Hospital "Hôpital de Mercy", Metz
  - Nancy University Hospita "Hôpitaux de Brabois", Nancy
  - Nantes University Hospital, Nantes
  - APHP "Hôpital Saint-Antoine", Paris
  - Rennes University Hospital, Rennes
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital "Hôpital Bretonneau", Tours

REFERENCES:
- [Derived] Zamagni E, Nanni C, Dozza L, Carlier T, Bailly C, Tacchetti P, Versari A, Chauvie S, Gallamini A, Gamberi B, Caillot D, Patriarca F, Macro M, Boccadoro M, Garderet L, Barbato S, Fanti S, Perrot A, Gay F, Sonneveld P, Karlin L, Cavo M, Bodet-Milin C, Moreau P, Kraeber-Bodere F. Standardization of 18F-FDG-PET/CT According to Deauville Criteria for Metabolic Complete Response Definition in Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2021 Jan 10;39(2):116-125. doi: 10.1200/JCO.20.00386. Epub 2020 Nov 5. PMID 33151787
- [Derived] Jamet B, Morvan L, Nanni C, Michaud AV, Bailly C, Chauvie S, Moreau P, Touzeau C, Zamagni E, Bodet-Milin C, Kraeber-Bodere F, Mateus D, Carlier T. Random survival forest to predict transplant-eligible newly diagnosed multiple myeloma outcome including FDG-PET radiomics: a combined analysis of two independent prospective European trials. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1005-1015. doi: 10.1007/s00259-020-05049-6. Epub 2020 Oct 2. PMID 33006656